CLINICAL TRIAL: NCT02583282
Title: A Study to Compare the Efficacy and Safety of Intrapleural Doxycycline Versus Iodopovidone for Performing Pleurodesis in Malignant Pleural Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: INT/IEC/2015/232
Record Dates: First submitted 2015-08-04; First posted 2015-10-22 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Experimental): Intrapleural doxycycline
  Interventions: Other: Doxycycline
- Iodopovidine (Active Comparator): Intrapleural iodopovidine
  Interventions: Other: Iodopovidine

INTERVENTIONS:
Other: Doxycycline — 500 mg of doxycycline will be dissolved in 50 ml of normal saline. The combination will then be instilled through the chest tube in the pleural cavity and the chest tube drain will be clamped for 4 hours.
  Arms: Doxycycline
Other: Iodopovidine — 20 ml of 10% betadine (Microshield, Johnson and Johnson, Solan, India) will be dissolved in 80 mL of normal saline. The combination will then be instilled through the chest tube in the pleural cavity and the chest tube drain will be clamped for 4 hours.
  Arms: Iodopovidine

SUMMARY:
Malignant pleural effusion (MPE) arises in advanced-stages of malignancies and frequently heralds a poor prognosis.If the underlying malignancy is chemo sensitive (e.g., small-cell carcinoma of lung & lymphoma), systemic chemotherapy may control the pleural effusion. Instilling of sclerosing agents into the pleural cavity (pleurodesis) is a common method for the management of MPE. According to a recent survey, tetracycline or its derivative (doxycycline) is the preferred agent for performing pleurodesis at many centers. In a previous study from the investigators' center, the investigators have demonstrated equal efficacy of iodopovidone in comparison to talc in inducing pleural symphysis. Also, iodopovidone has been postulated to have anti-neoplastic effects and hence may help in reducing the drain output. Apart from these benefits iodopovidone is easily available and is cost effective. The investigators believe that iodopovidone will have better efficacy than doxycycline in inducing pleurodesis in malignant pleural effusion.

DETAILED DESCRIPTION:
Introduction & Review of literature Malignant pleural effusion (MPE) arises in advanced-stages of malignancies and frequently heralds a poor prognosis. Most patients with MPE are symptomatic. The most common symptom is exertional dyspnea. Most patients undergo chemotherapy or local treatments to palliate symptoms such as dyspnea, cough & chest pain, to improve quality of life. If the underlying malignancy is chemo sensitive (e.g., small-cell carcinoma of lung & lymphoma), systemic chemotherapy may control the pleural effusion.1 However, when pleural effusion persists or reaccumulates after chemotherapy, the management of refractory MPE includes local therapeutic methods such as thoracentesis, pleurodesis, pleurectomy, or pleuroperitoneal shunting. Instilling of sclerosing agents into the pleural cavity (pleurodesis) is a common method for the management of MPE. For several years, various agents such as anti-neoplastics (e.g., nitrogen mustard, bleomycin), tetracycline derivatives, talc, erythromycin, silver nitrate, and povidone-iodine have been injected into the pleural cavity to create pleurodesis.

According to a recent survey, tetracycline or its derivative (doxycycline) is the preferred agent for performing pleurodesis at many centers.7 However, intravenous preparation of doxycycline is not freely available and also induces severe inflammation in the pleura that results in severe chest pain and discomfort to the patient. In a previous study from the investigators' center, the investigators have demonstrated equal efficacy of iodopovidine in comparison to talc in inducing pleural symphysis.8 Also, iodopovidine has been postulated to have anti-neoplastic effects and hence may help in reducing the drain output. Apart from these benefits iodopovidine is easily available and is cost effective. The investigators believe that iodopovidone will have better efficacy than doxycycline in inducing pleurodesis in malignant pleural effusion.

Study hypothesis In patients with malignant pleural effusion, pleurodesis with intrapleural instillation of iodopovidone will have better efficacy in comparison with doxycycline.

Methods

Study design: This will be a randomized double blind study conducted in the Department of Pulmonary Medicine, PGIMER, Chandigarh.

Selection of cases: A total of 100 consecutive patients of malignant pleural effusion will be enrolled in the study. Patients will be equally randomized to undergo pleurodesis, either with intrapleural iodopovidone or intrapleural doxycycline. A written informed consent will be taken from all the patients participating in the present study

Randomization: Patient will be randomized 1:1 to undergo pleurodesis either by instillation of intrapleural iodopovidone or intrapleural doxycycline. The randomization sequence will be computer generated. The sequence generated will be kept in a sealed opaque envelope and will be opened at the time of procedure

Procedure: A chest tube (24-28 F) will be inserted through the fifth intercostal space in the mid-axillary line, to achieve complete drainage of the effusion and/or complete lung expansion. In case of large effusions, drainage will be spread over 24-48 h to prevent re-expansion pulmonary oedema. Pleurodesis will be performed when the daily drainage output will decrease to <150 mL/day and chest radiograph demonstrates apposition of pleural surfaces. In cases of pneumothorax, complete lung expansion and absence of any air leaks will be confirmed before instillation of the chemical agent. A chest radiograph will be performed to confirm complete re-expansion. Normal saline solution (50 mL) containing lignocaine (2 mg/kg ideal body weight) will be infused through the chest tube. Simultaneously, tramadol (100 mg) will be administered intravenously for analgesia. After 15 minutes pleurodesis will be performed either by instillation of doxycycline or by iodopovidone.

Doxycycline: 500 mg of doxycycline will be dissolved in 50 ml of normal saline. The combination will then be instilled through the chest tube in the pleural cavity and the chest tube drain will be clamped for 4 hours.

Iodopovidone: 20 ml of 10% betadine (Microshield, Johnson and Johnson, Solan, India) will be dissolved in 80 mL of normal saline. The combination will then be instilled through the chest tube in the pleural cavity and the chest tube drain will be clamped for 4 hours.

The chest tube will be flushed with 50 mL of normal saline after instillation of study drug (doxycycline or iodopovidone).

Endpoint: The chest tube will be removed if the drainage output is less than 100mL of pleural fluid and there is complete lung re-expansion with no residual pneumothorax on chest radiograph. Pulse, blood pressure, respiratory rate and temperature will be measured before and every 30 minutes after the procedure for 6 hours. Chest pain after pleurodesis will be recorded on a visual analogue scale (VAS) of 0-100 mm. Patients will be given additional intravenous tramadol (50 mg) on an as-needed basis after the procedure. Any complications related to the procedure will be recorded. Complications such as hypotension, fever, acute respiratory failure and empyema will be noted. Patients will be followed up at 1 week, at 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* recurrent symptomatic malignant pleural effusion, with subjective improvement of dyspnea following thoracentesis

Exclusion Criteria:

* history of any allergy to iodine or doxycycline
* history of thyroid disorders
* failure of lung expansion after insertion of intercostal tube (trapped lung)
* presence of air leaks
* advanced malignancy with limited predicted life expectancy (<30 days)
* failure to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Complete success | 30 days
  long-term relief of symptoms related to the effusion, with absence of re-accumulation of fluid on chest radiograph at 30 days
Partial success | 30 days
  diminution of dyspnea related to the effusion, with only partial reaccumulation of fluid and no requirement for therapeutic thoracentesis
Failed pleurodesis | 30 days
  reaccumulation of pleural fluid requiring therapeutic thoracentesis, persistence of drainage output >250mL/day requiring repeat procedure, lack of success requiring surgical intervention

SECONDARY OUTCOMES:
Time to pleurodesis | 1 week
  interval between instillation of the agent and removal of the chest tube

CONTACTS AND LOCATIONS:
Locations (1):
- Bronchoscopy suite, PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Damaraju V, Sehgal IS, Muthu V, Prasad KT, Dhooria S, Aggarwal AN, Agarwal R. Efficacy and safety of doxycycline versus iodopovidone for pleurodesis through an intercostal tube in malignant pleural effusions: a randomized trial. Support Care Cancer. 2023 Jul 10;31(8):454. doi: 10.1007/s00520-023-07932-y. PMID 37428348